CLINICAL TRIAL: NCT05166538
Title: Dual Antiplatelet Therapy in Patients With Clopidogrel Resistance Following Off-Pump Coronary Artery Bypass: Prospective, Randomized Controlled Trial
Brief Title: Dual Antiplatelet Therapy in Patients With Clopidogrel Resistance Following Off-Pump Coronary Artery Bypass
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-2374-001
Record Dates: First submitted 2021-08-20; First posted 2021-12-22 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: Multi Vessel Coronary Artery Disease
Keywords: Antiplatelets; Coronary artery bypass surgery
MeSH Terms: interventions — Ticagrelor; Clopidogrel

STUDY DESIGN:
Intervention Model Description: Postoperative cardiac surgery, patients were randomized to receive ticagrelor or clopidogrel (n=102), respectively. The selected agent was applied in the operating room.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ticagrelor (Experimental)
  Interventions: Drug: Ticagrelor
- Clopidogrel (Active Comparator)
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Ticagrelor — direct-acting oral P2Y12-receptor antagonist
  Other Names: brilinta
  Arms: Ticagrelor
Drug: Clopidogrel — platelet aggregation inhibitor
  Other Names: plavix
  Arms: Clopidogrel

SUMMARY:
Ticagrelor, a direct-acting oral P2Y12-receptor antagonist, provides greater and more consistent platelet inhibition than clopidogrel. This study aimed to compare outcomes of ticagrelor plus aspirin versus clopidogrel plus aspirin 1 year after off-pump coronary artery bypass grafting (OPCAB) in patients with clopidogrel resistance.

DETAILED DESCRIPTION:
Between November 2014 and November 2020, 1739 patients underwent OPCAB. Aspirin (100mg daily) and clopidogrel (75mg daily) were administered beginning at aday 1 after surgery. On the 7th postoperative day, the clopidogrel resistance was evaluated by point-of-care assay. Among them, the patients had clopidogrel resistance were enrolled in this study. Investigators divide them into two groups [A: ticagrelor, B; clopidogrel]. Primary endpoint was all-cause of mortality 1 year after OPCAB. Secondary endpoint included major adverse cardiovascular events (MACE: cardiac death, myocardial infarction, or stroke). Multivariate Cox regression was used to evaluate predictors of end points.

ELIGIBILITY:
Inclusion Criteria:

1. patients aged 19 years or older
2. undergoing elective OPCAB surgery with multi-vessel coronary artery disease.

Exclusion Criteria:

1) patient had aspirin resistance

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Early graft patency | 1 year after OPCAB
  graft occlusion rate diagnosed by CT exam, at follow-up angiography, grafts were evaluated by use of the usual definition of patency and were assessed for FitzGibbon patency with the A, B, and O classification system in which FitzGibbon A is an excellent/unimpaired graft, Bis an impaired graft with a stenosis >50% reducing the caliber of the graft to <50% of the target artery diameter, and O is a completely occluded graft.

SECONDARY OUTCOMES:
degree of resistance | 7 day after surgery
  Platelet reactivity was assayed using the VeriofyNowP2Y12 assay (Accumetrics Inc, San Diego, CA) which is a cartridge-based assay that specifically measures the direct effects of clopidogrel on the platelet P2Y12 receptor. The results are expressed as P2Y12 reaction units (PRUs) for clopidogrel. The cut-off PRU value was 188 PRU and the details were described previous study.
Number of patients with resistance with clopidogrel as assessed by VeriofyNowP2Y12 assay | 7 day after surgery
  The cut-off PRU value was 188 PRU
Mediastinal Bleeding | up to 4 weeks
  total drainage counts (ml) from median tubes
Total hospital day from admission to discharge | up to 4 weeks
rate of postoperative stroke of myocardial infarction | Participants will be followed during 1 years from operation
rate of postoperative morbidity/ mortality | Participants will be followed during 5 years from operation

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Yonsei University Health System, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Varma PK, Ahmed H, Krishna N, Jose R, Gopal K, Mathew OP, Jayant A. Bleeding complications after dual antiplatelet therapy with ticagrelor versus dual antiplatelet therapy with clopidogrel-a propensity-matched comparative study of two antiplatelet regimes in off-pump coronary artery bypass grafting. Indian J Thorac Cardiovasc Surg. 2021 Jan;37(1):27-37. doi: 10.1007/s12055-020-01052-6. Epub 2020 Oct 7. PMID 33442205